CLINICAL TRIAL: NCT05376020
Title: A Randomised Control Clinical Trial Investigating the Effect of Osseodensification on Implant Stability and Marginal Bone Levels
Brief Title: Osseodensification and Dental Implant Stability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Ioanna Politi, Principal Investigator, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPoliti
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Osseointegration; Osseodensification

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Densah Burs (Experimental): Intervention Group
  Interventions: Device: Densah Burs
- Conventional Burs (Active Comparator): Control Group
  Interventions: Device: Conventional Burs

INTERVENTIONS:
Device: Densah Burs — Densah Burs will be used in the intervention group
  Arms: Densah Burs
Device: Conventional Burs — Conventional Burs will be used in the control group
  Arms: Conventional Burs

SUMMARY:
Osseointegration refers to the formation of a structural and functional bone-to-implant interface, without the interposition of soft tissue. Successful osseointegration will provide long term success for the dental implant. Primary implant stability, is the mechanical stability between bone and the implant at the time of insertion and is key to initiate a successful osseointegration.

Both primary implant stability and osseointegration are affected by the density of the bone where the implant is placed. A relatively new technique known as osseodensification (OD) has been developed and uses specially designed burs (Densah burs). Compared to conventional drills (CD) that remove bone (subtractive drilling) these burs are designed so that they can rotate in a counterclockwise (CCW) (non subtractive) direction which allows bone to be preserved and compacted into the wall of the osteotomy site. These drills therefore theoretically maintain bone volume which then creates higher bone density and bone to implant contact allowing better implant primary stability.

This study will be a randomised control trial comparing OD to CD with regards to implant stability and bone levels. Considering the increased cost of OD, available literature must support a significant clinical benefit of OD over CD to consider them for clinical use. This study will aim to reinforce available clinical research and address some of the limitations of the current evidence to aid clinicians in making an evidenced-based decision on the use of OD when poor bone density could compromise implant success.

ELIGIBILITY:
Inclusion Criteria:

Patient Level

* Male or Female, 18 years old or over
* Capacity to provide informed consent
* Willing to comply with study appointment schedule Willing to maintain a diary of symptoms
* Planned for provision of dental implant(s) at Dublin Dental University Hospital

Site Level

* Location: maxilla
* Sufficient bone volume for implant placement without the need for bone graft/augmentation; alveolar ridge of minimum 6mm width for standard implants (implant diameter 4mm) and of minimum 7mm for wider implants (implant diameter 5mm)

Exclusion Criteria:

Patient Level

* Plaque score >20%
* Bleeding score >20%
* Tobacco smoking
* Uncontrolled systemic disease
* Use of systemic medications with an expected impact on bone healing (e.g. bisphosphonates)
* Pregnancy or lactation
* Lack of capacity to give an informed consent

Site Level

* Location: mandible
* Insufficient bone volume for implant placement, requiring bone graft/augmentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-05-13 (Estimated); Primary Completion 2024-05-13 (Estimated); Study Completion 2024-05-13 (Estimated)

PRIMARY OUTCOMES:
Implant Stability | During procedure (implant placement)
  Implant stability Quotient (ISQ) will be measured using magnetic resonance frequency analysis (MRFA) - the device is called OSSTELL. A transducer is attached to the implant and brought to vibration by magnetic pulses from the probe of the Osstell device which makes the implant vibrate. The implant's resistance to vibration is expressed as the ISQ value. High vibration frequency signifies high implant stability.
Implant Stability | At time of second stage implant surgery (3 months)
  Implant stability Quotient (ISQ) will be measured using magnetic resonance frequency analysis (MRFA) - the device is called OSSTELL. A transducer is attached to the implant and brought to vibration by magnetic pulses from the probe of the Osstell device which makes the implant vibrate. The implant's resistance to vibration is expressed as the ISQ value. High vibration frequency signifies high implant stability.
Implant Stability | At implant restoration (5 months)
  Implant stability Quotient (ISQ) will be measured using magnetic resonance frequency analysis (MRFA) - the device is called OSSTELL. A transducer is attached to the implant and brought to vibration by magnetic pulses from the probe of the Osstell device which makes the implant vibrate. The implant's resistance to vibration is expressed as the ISQ value. High vibration frequency signifies high implant stability.

SECONDARY OUTCOMES:
Insertion torque | During procedure (implant placement)
  Insertion torque of implant will be measured using standard torque wrench
Marginal bone levels | During procedure (implant placement)
  Will be measured clinically using a periodontal probe and radiographically
Marginal bone levels | At time of second stage implant surgery (3 months)
  Will be measured clinically using a periodontal probe
Marginal bone levels | At implant restoration (5 months)
  Will be measured clinically using a periodontal probe and radiographically

CONTACTS AND LOCATIONS:
Locations (1):
- Dublin Dental Hospital/Trinity College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Politi I, Honari B, Winning L, Polyzois I. The Effect of Osseodensification on Implant Stability and Marginal Bone Levels: A Randomized Control Clinical Trial. Clin Exp Dent Res. 2025 Feb;11(1):e70126. doi: 10.1002/cre2.70126. PMID 40205940